CLINICAL TRIAL: NCT07375914
Title: Comprehensive Biopsychosocial Approach for Acute Low Back Pain Management in the Emergency Department: a Stepped-wedge Cluster-randomized Clinical Trial
Acronym: CALM-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP251083; IDRCB: 2025-A01588-41 (Other: ANSM)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-traumatic Low Back Pain
Keywords: Emergency medicine; Acute Low back pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual care - Standard care for acute non-specific low back pain at clinician's discretion
- Intervention group (Experimental): Biopsychosocial approach
  Interventions: Other: Biopsychosocial intervention

INTERVENTIONS:
Other: Biopsychosocial intervention — The biopsychosocial intervention consists of a structured program implemented in participating emergency departments. It includes a standardized 3-hour online training session for physicians covering evidence-based management of acute low back pain, rational pharmacological use, promotion of physical activity, and consideration of psychosocial factors. A summary sheet will be given with key recommendations during the period. For patients, short educational materials provide information on typical recovery, self-management strategies, and appropriate follow-up. The intervention is introduced sequentially across 12 centers according to a stepped-wedge randomization schedule, with each site moving from control to intervention while maintaining standard emergency care.
  Arms: Intervention group

SUMMARY:
Acute low back pain, the second leading cause of medical consultations in France, poses a major public health challenge, particularly because of its high risk of progressing to chronic low back pain-the leading cause worldwide of years lived with disability. Pharmacological treatments such as paracetamol, opioids, non-steroidal anti-inflammatory drugs (NSAIDs) and muscle relaxants show limited benefit in terms of pain intensity or functional disability. Non-pharmacological treatments, including exercise therapy and psychological support, show promising results but remain hampered by methodological biases and small sample sizes.

A biopsychosocial approach that combines pharmacological treatments, physical therapy, psychological support and social interventions has demonstrated moderate improvements in pain and function for chronic low back pain but remains insufficiently studied for acute presentations. French guidelines advocate a combined strategy involving paracetamol, NSAIDs, physical activity and psychosocial risk assessment. However, a French multicentre retrospective study highlighted marked heterogeneity in clinical practice, along with a low adoption rate (<10 %) of these recommendations in emergency departments, underscoring the need to strengthen adherence to evidence-based management strategies. We hypothesise that a multimodal intervention targeting physicians (guideline reminders) and patients (information on disease progression and multidisciplinary care plans), to enable the systematic implementation of all aspects of a biopsychosocial approach in emergency departments, could reduce short-term pain and disability in patients with acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 55 presenting to a participating emergency department, and
* Presenting with acute non-traumatic low back pain, newly developed or worsened within the past 7 days.
* Moderate to severe pain, defined as a score of ≥4 on a 0-10 numerical rating scale.
* Provision of informed consent after being given the information sheet.
* Patients covered by social security (excluding AME).

Exclusion Criteria:

* Presence of a 'red flag' according to HAS guidelines, including: motor neurological deficit or cauda equina syndrome, non-mechanical pain, trauma, active neoplastic disease or history of inflammatory rheumatism, suspected osteoarticular infection, recent spinal surgery with worsening symptoms, suspected acute vascular pathology, prolonged use of medications or corticosteroids, significant structural spinal deformity, or deterioration of general health.
* Inability to attend the 3-month follow-up.
* Poor command of French.
* Patient under guardianship/curatorship or deprived of liberty.
* Pregnant or breastfeeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 782 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain Interference Score at 7 days | 7 days
  Pain interference score at 7 days, assessed using the Pain Interference subscale of the Brief Pain Inventory - Short Form (BPI-SF). The score is calculated as the mean of 7 items (each rated 0-10) and reported on a 0-100 scale

SECONDARY OUTCOMES:
Pain intensity at 7 days, measured by the BPI SF intensity score. | 7 days
Number of pain-free days after the emergency department visit | 7 days
  Number of days with BPI intensity at 0
Total amount of opioids consumed | 7 days and 3 months
  Proportion of patients pain-free at 7 days and at 3 months : Total amount of opioids consumed at 7 days and at 3 months (in morphine equivalent).
Number of days off work | 7 days and 3 months.
  Number of days off work at 7 days and at 3 months.
Functional disability | 3 months
  Functional disability at 3 months, measured using the Roland-Morris Disability Questionnaire.
Patient satisfaction and quality of life | 3 months
  Patient satisfaction and quality of life at 3 months, assessed using the EQ-5D-5L
Number of X-rays, CT scans, and MRI scans of the spine performed | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Héloïse BANNELIER, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No